CLINICAL TRIAL: NCT04322279
Title: Factors Associated With a Positive SARS-CoV-2 Serology in Contact Subjects at High/Moderate Risk of Coronavirus SARS-CoV-2 Infection. (CoV-CONTACT-SERO)
Brief Title: Factors Associated With a Positive SARS-CoV-2 Serology in Contact Subjects at High/Moderate Risk of Coronavirus SARS-CoV-2 Infection. COVID-19.
Status: Terminated | Type: Observational
Why Stopped: no topics to include
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-16; 2020-A00609-30 (Registry Identifier: RCB-ID)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Coronavirus
Keywords: contact subject; high/moderate risk of transmission
MeSH Terms: conditions — Coronavirus Infections | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serology — SARS-CoV-2 serology
Genetic: Sequencing — Whole exome sequencing

SUMMARY:
In December 2019, a pneumonia due to a novel coronavirus (SARS-CoV-2) emerged in the city of Wuhan, in China. In a few weeks, the number of confirmed cases of SARS-CoV-2 infection has dramatically increased, with almost 150'000 cases and more than 6'000 reported deaths on March, 16th 2020.

Little is known on the rate of human-to-human transmission of this new coronavirus SARS-CoV-2 in the community and within the hospital.

Depending on the country, contact subjects considered to be at high or moderate risk of SARS-CoV-2 are, either isolated at home for a period of time defined by the health authorities or, on the contrary, continue their professional activity on the condition that they adopt measures to prevent transmission to those around them. In most European countries, healthcare workers adopt this second option. In all cases, it is most often recommended that contact persons monitor their state of health and communicate it to the persons dedicated to this action.

Whether such subjects become spreaders of the virus is not known, nor is the proportion of viral spreader who will develop a symptomatic infection.

In this study, we aim to evaluate the virological and clinical outcomes of subjects following a contact at high/moderate risk of SARS-CoV-2 acquisition, in community-subjects and/or healthcare workers.

The study population is represented by all subjects who had a contact with laboratory-confirmed SARS-CoV-2 cases and whose contact was considered to be at high/moderate risk of SARS-CoV-2 acquisition.

This include both children and adult subjects, subject without social security, and healthcare workers.

DETAILED DESCRIPTION:
Procedures added by the research:

Blood sampling for determination of the presence of SARS-CoV-2 type M immunoglobulins or type G immunoglobulins.

Blood sampling for whole exome sequencing

ELIGIBILITY:
Inclusion Criteria:

* High/moderate risk contact with a laboratory-confirmed SARS-CoV-2 case;
* Within the 14 days following the last contact with a laboratory-confirmed SARS-CoV-2 case;
* Obtaining informed consent.

Exclusion Criteria:

* Subject included in the CoV-CONTACT study
* Subject deprived of freedom
* Subject under a legal protective measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is represented by all subjects who had a contact with laboratory-confirmed SARS-CoV-2 cases and whose contact was considered to be at high/moderate risk of SARS-CoV-2 acquisition.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with SARS-CoV-2 positive serology at day 30 following the last high/moderate risk contact with a laboratory-confirmed SARS-CoV-2 case. | 30 days (+/-7)
  Positive serology defined as the presence of SARS-CoV-2 IgM or IgG and assessed by ELISA, microneutralisation assay

SECONDARY OUTCOMES:
Factors associated with a SARS-CoV-2 positive serology at day 30 (+/-7); | 30 days (+/-7)
  Positive serology defined as the presence of SARS-CoV-2 IgM or IgG and assessed by ELISA, microneutralisation assay
Time (days) between the first positive SARS-CoV-2 serology and the first negative SARS-CoV-2 serology. | 365 days (+/-30)
  ELISA, microneutralisation assay

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DUVAL, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (16):
- France (15):
  - Service de maladies infectieuses et tropicales Hôpital Jean Minjoz CHRU Besançon, Besançon
  - Service des Maladies infectieuses et tropicales, Pôle Spécialités médicales, CHU Pellegrin, Bordeaux
  - Service des maladies infectieuses Hôpital Gabriel Montpied CHU de Clermont Ferrand, Clermont-Ferrand
  - Centre d'investigation clinique 1432 Hôpital François Mitterrand CHU Bourgogne, Dijon
  - Centre d'investigation clinique 1406 CHU Grenoble, Grenoble
  - Centre d'Investigation Clinique 1403 -CHU Lille, Lille
  - Centre d'Investigation Clinique Hôpital Saint Louis, Paris
  - Centre d'investigation Clinique 1425, Hôpital Bichat Claude Bernard, Paris
  - Hôpital Cochin CIC 1417 Bâtiment Lavoisier, Paris
  - Centre d'investigation clinique 1414 Service de Pharmacologie clinique CHU Rennes Hôpital Pontchaillou, Rennes
  - Centre Hospitalier Félix Guyon Ile de la Réunion CHU nord, Saint-Denis
  - Département maladie infectieux CHU Saint Etienne, Saint-Etienne
  - Centre d'Investigation Clinique Ile de la Réunion CHU sud, Saint-Pierre
  - Centre Investigation Clinique 1415 CHRU Tours - Hôpital Bretonneau, Tours
  - Centre Investigation Clinique 1433 CHRU de NANCY, Vandœuvre-lès-Nancy
- Service de Maladies infectieuses et tropicales Centre hospitalier, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided